CLINICAL TRIAL: NCT02231710
Title: A Study Evaluating BPX-501 T Cells and AP1903 for Prevention of Graft Versus Host Disease (GVHD) After Haploidentical, Related, T Cell-Depleted Hematopoietic Cell Transplantation for Non-Malignant Diseases
Brief Title: Safety Study of Gene Modified Donor T Cell Infusion After Stem Cell Transplant for Non-Malignant Diseases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to lack of enrollment and changes to the sponsor development portfolio
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-003
Expanded Access: NCT03639844 (No longer available)
Record Dates: First submitted 2014-08-28; First posted 2014-09-04 (Estimated); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-09

CONDITIONS: Primary Immune Deficiency Disorders; Hemophagocytic Lymphohistiocytosis; Inherited Bone Marrow Failure Syndrome; Hemoglobinopathies; Metabolic Disorders
Keywords: Severe Combined Immune Deficiency; Congenital T-cell Defect; Congenital T-cell Deficiency; Chronic Granulomatous Disease; Shwachman Diamond Syndrome; Diamond Blackfan Anemia; Dyskeratosis Congenita; Fanconi Anemia; Sickle Cell Disease; Thalassemia; Mucopolysaccharidosis; Sphingolipidoses
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Lymphohistiocytosis, Hemophagocytic; Congenital Bone Marrow Failure Syndromes; Hemoglobinopathies; Metabolic Diseases; Severe Combined Immunodeficiency; Granulomatous Disease, Chronic; Shwachman-Diamond Syndrome; Anemia, Diamond-Blackfan; Dyskeratosis Congenita; Fanconi Anemia; Anemia, Sickle Cell; Thalassemia; Mucopolysaccharidoses; Sphingolipidoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BPX-501 and Rimiducid (Experimental): Single administration of BPX-501 T cells post partially-mismatched, related T cell depleted HCT followed by Rimiducid infusion on day 7
  Interventions: Biological: BPX-501 and Rimiducid

INTERVENTIONS:
Biological: BPX-501 and Rimiducid — Single administration of BPX-501 T cells post partially-mismatched, related T cell depleted HCT followed by Rimiducid infusion on day 7

SUMMARY:
The purpose of this study is to determine a safe dose of BPX-501 gene modified T cells infused after a haplo-identical stem cell transplant to facilitate engraftment and the safety of Rimiducid (AP1903) on day 7 to prevent GVHD.

DETAILED DESCRIPTION:
This is a single arm dose finding study evaluating the safety and efficacy of a BPX 501 infusion (T cells genetically modified with the inducible Caspase 9 suicide gene) of 3x10E6 to 1X10E7 cells/kg followed by a Rimiducid infusion on day 7 after a partially mismatched, related, T cell-depleted hematopoietic cell transplantation (HCT) in patients with non-malignant diseases. The purpose of this clinical trial is to determine the dose of BPX 501 T cell infusion with subsequent planned infusion of Rimiducid which can facilitate engraftment and prevent the occurrence of GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must meet eligibility criteria for allogeneic transplantation
2. Lack of suitable conventional donor (10/10 allele matched related or unrelated donor) or presence of rapidly progressive disease not permitting time to identify an unrelated donor
3. Males or females
4. Age < 55 years old and > 4 months
5. Diagnosis of a nonmalignant disorder considered treatable by HCT.
6. HLA typing will be performed at high resolution (allele level) for the HLA-A, -B, Cw, DRBl, and DQB1 loci.

   i. A minimum match of 5/10 is required. ii. The donor and recipient must be identical, as determined by high resolution typing, in at least one allele of each of the following
7. If capable of reproduction, patient must agree to use contraception or abstinence to prevent pregnancy during the first year of enrollment and treatment.
8. Informed consent signed by patient (if ≥18 years old) or parent/guardian (if <18 years old).
9. Fanconi anemia patients ONLY i) Patients must meet one of the following criteria to be eligible for this study:

   1. Any patient with Fanconi anemia and bone marrow failure involving 2 of the following 3 lineages: granulocyte count <0.5 x 109/L, platelet count <20 x 109/L, or hemoglobin <8 g/dL.
   2. Any patient with Fanconi anemia who requires red blood cell or platelet transfusions because of marrow failure
   3. Any patient with Fanconi anemia who has a life-threatening bone marrow failure involving a single hematopoietic lineage.

Exclusion Criteria:

1. Serious organ dysfunction
2. Pregnant or breast-feeding
3. Evidence of HIV infection
4. Bovine product allergy
5. Patients with an active infectious disease
6. Patients with Fanconi anemia with AML/MDS.

Ages: 4 Months to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bellicum Pharmaceuticals Senior Director, Study Director — Clinical Development
Locations (1):
- Fred Hutchinson Cancer ResearchCenter, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BPX-501 and Rimiducid: Single administration of BPX-501 T cells (5 x 10^6 cell/kg), post partially-mismatched, related T cell depleted HCT followed by Rimiducid infusion on day 7
  BPX-501 and Rimiducid: Single administration of BPX-501 T cells post partially-mismatched, related T cell depleted HCT followed by Rimiducid infusion on day 7
  NOTE: This study enrolled a single patient and was terminated early due to lack of enrolment
Period: Overall Study
Arm/Group | BPX-501 and Rimiducid
Started | 1
Completed | 0
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | BPX-501 and Rimiducid
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 12 [12 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1
sickle cell disease [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: To determine the safety (as defined by non-responsive Grade III-IV GVHD to rimiducid) of HCT with HLA-haploidentical CD34+ selected peripheral blood stem cell (PBSC) grafts and BPX 501 T cells followed by scheduled rimiducid infusion on Day 7.
  this outcome measure is reported as number of patients who experienced the AE of Grade III-IV GVHD that was not non-responsive to rimiducid (safety switch) administration.
Time Frame: 24 months
Population: One subject was dosed with 5 x 106 cells of BPX-501 T cells and 0.4 mg/kg of rimiducid on Day 7. No efficacy data was gathered for this patient and patient was withdrawn from the Study by investigator's physician. The study was terminated early by Sponsor due to lack of enrolment
Arm/Group | BPX-501 and Rimiducid
Number analyzed (Participants) | 0

2. Primary Outcome: Engraftment
Description: Determine the engraftment rate (defined as >50% donor CD3 chimerism) on day 28 after HCT with HLA-haploidentical CD34+ selected PBSC grafts per dose cohort of BPX 501 T cells followed by Rimiducid infusion on Day 7.
  NOTE: only one patient was enrolled who received the dose of 5x 10^6cell/kg dose of BPX-501
Time Frame: Day 28
Population: as for outcome 1
Arm/Group | BPX-501 and Rimiducid
Number analyzed (Participants) | 0

3. Secondary Outcome: GvHD
Description: To determine the incidence and severity of acute and chronic GVHD
Time Frame: Month 24
Reporting Status: Not Posted

4. Secondary Outcome: Immune Reconstitution
Description: Measure immune reconstitution
Time Frame: Month 24
Reporting Status: Not Posted

5. Secondary Outcome: Infection Rates
Description: Determine the risk for severe infections
Time Frame: Day 200
Reporting Status: Not Posted

6. Secondary Outcome: Graft Rejection
Description: Incidence of graft rejection
Time Frame: Month 24
Reporting Status: Not Posted

7. Secondary Outcome: Rimiducid Activity
Description: Time to resolution of acute and chronic GvHD following administration of Rimiducid
Time Frame: Month 24
Reporting Status: Not Posted

8. Secondary Outcome: High Grade Toxicity
Description: Rate of high grade toxicity
Time Frame: Month 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: was intended for 24 months
Description: Adverse events were collected via questioning or subject-reporting and were subsequently coded in tabular form using the MedDRA Version 21.0 adverse event dictionary and CTCAE designations (in lieu of Grade 1-4 classification)
Groups:
- BPX-501 and Rimiducid: Single administration of BPX-501 T cells (5 x 10^6 cell/kg), post partially-mismatched, related T cell depleted HCT followed by Rimiducid infusion on day 7
  BPX-501 and Rimiducid: Single administration of BPX-501 T cells post partially-mismatched, related T cell depleted HCT followed by Rimiducid infusion on day 7
  NOTE: This study enrolled a single patient who discontinued the study due to investigating physicians decision. The study was terminated early due to lack of enrolment.
Arm/Group | BPX-501 and Rimiducid
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPX-501 and Rimiducid (N=1)
haemolysis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPX-501 and Rimiducid (N=1)
Platelet Count Decreased (Investigations) | 1 (22)
Haematocrit Decreased (Investigations) | 1 (8)
Activated Partial Thromboplastin Time abnormality (Investigations) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT02231710/Prot_000.pdf